CLINICAL TRIAL: NCT01380340
Title: Study of the Effects of a New Concept of Early Intervention on the Driving Cessation, Mental Health, and Quality of Life of Senior Drivers
Brief Title: Seniors Driving Cessation Early Intervention Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Jane Rodwell, Occupational Therapist, Fraser Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FHREB# 2011-051
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Depression; Quality of Life
Keywords: Seniors; Driving; Group work
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seniors early intervention driving group (Experimental): The seniors early intervention driving group is for seniors who have been identified by professionals as having to face changes to their driving status. It involves activities such as change strategies, positive psychology approaches and topic based discussion designed to mitigate the health and quality of life effects of driving regulation and cessation.
  Interventions: Other: Seniors Early Intervention Planning and Discussion.
- Matched comparison group (No Intervention): The subjects will be recruited from a parallel service and will be paired with similar subjects in the experimental group.

INTERVENTIONS:
Other: Seniors Early Intervention Planning and Discussion. — The seniors early intervention driving group is for seniors who have been identified by professionals as having to face changes to their driving status. It involves activities such as change strategies, positive psychology approaches and topic based discussion designed to mitigate the health and quality of life effects of driving regulation and cessation.
  Arms: Seniors early intervention driving group

SUMMARY:
This study will investigate the effects of a new form of early intervention for senior drivers who are at risk of changes to their driving status. The early intervention consists of group activities involving planning and professionally facilitated discussion.

There are three main research hypotheses for this study. Firstly, it is hypothesised that early intervention, in the form of the information and planning group, will not be associated with either increases or decreases in driving assessment failure or driving cessation. Secondly, it is hypothesised that early intervention will be associated with patterns of reduced depression and less persistent negative mood states. Thirdly, it is hypothesised that early intervention will be associated with patterns of sustained levels of important quality of life indicators such as community participation and social relationships.

DETAILED DESCRIPTION:
Study Protocol Summary:

This Canadian, British Columbian study, in the Fraser Health Authority region will involve seniors who have been referred to two Specialized Seniors Clinics (SSC) and have been flagged by clinicians for report to the Office of the Superintendent of Motor Vehicles (OSMV) for a driving assessment. At the White Rock/South Surrey (WR/SS) SSC,British Columbia (BC),10 subjects will be invited to participate in an information and planning group. Ten additional subjects from New Westminster (NW), BC SSC, will be matched with group participants. Each subject will be interviewed by an occupational therapist during which time the Geriatric Depression Scale (GDS)and an abbreviated version of the World Health Organization Seniors Quality of Life Brief Questionnaire (WHOQOL-BREF) will be administered. Each subject will be contacted by phone bi-monthly for 10 months and the tests will be re-administered. During the phone calls additional information about each senior's driving status and driving patterns will be collected.

Background Information:

This type of early intervention has not previously been researched or made available. Research has shown that seniors who lose their driving license are at increased risk of depression and social isolation. The PI research that preceded this study demonstrated that seniors who had experienced enforced loss of their driving license often showed long-term negative emotions such as anger and bitterness coupled with a sense of injustice.

Purpose of Study The purpose of the study is to explore evidence of possible effects of an early intervention group in the areas of mood, quality of life and community access.

Justification for Study:

An important justification for this study is to examine the effects of a new concept of early intervention. Previous forms of intervention with existing senior drivers prior to assessment have involved activities such as public education and mature driver workshops. These have been evaluated in terms of the growth of knowledge and driving safety. In contrast, the new concept of early intervention involves activities such as group change strategies, positive psychology approaches and topic based discussion designed to mitigate the health and quality of life effects of regulation and cessation. In researching this new concept of early intervention, this project is intended to open up a new field for research. It will provide evidence of what effects can follow from early intervention and will indicate topics to be explored in subsequent research. In addition it will establish a model for the longitudinal research of senior drivers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be invited to participate in the study if they have been referred to the SSC at the start of the study and have a medical condition which is believed to have a potential impact on their driving. They will be living in the community at the time of their referral and they will also be driving their vehicle at that point in time.

Exclusion Criteria:

* Subjects do not qualify to participate in this study if they are not holding a current driving license at the time of recruitment and if they do not have a medical condition that effects their ability to drive.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Geriatric Depression Scale | 10 months
  The Geriatric Depression Scale (short form)is a well researched, standardized measure of depressive symptoms.It will be administered at the beginning and at the end of the study.
World Health Organization Quality of Life Measure (Brief) | 10 months
  The WHOQOL-BREF is a short version of the quality of life measure for seniors developed by the World Health Organization. It will be administered at the start and end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Rodwell, MA, Principal Investigator — Fraser Health Authority
Locations (2):
- Canada (2):
  - New Westminster Specialized Seniors Clinic, New Westminster, British Columbia
  - White Rock Specialized Seniors Clinic, White Rock, British Columbia